CLINICAL TRIAL: NCT01373918
Title: Low Dose Parenteral Fat for the Prevention of Parenteral Nutrition Associated Cholestasis in Neonates With Congenital/Acquired Gastrointestinal Disorders
Brief Title: Low Dose Fat for the Prevention of Liver Disease in Babies With Gastrointestinal Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to slow enrollment.
Sponsor: University of California, Los Angeles (Other)
Collaborators: St. Louis University (Other)
Responsible Party: Principal Investigator, Kara L. Calkins, MD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-001714
Record Dates: First submitted 2011-06-06; First posted 2011-06-15 (Estimated); Results first posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Cholestasis
Keywords: cholestasis; neonates; parenteral nutrition; gastrointestinal disorders
MeSH Terms: conditions — Cholestasis; Hyperphagia; Gastrointestinal Diseases | interventions — soybean oil, phospholipid emulsion; Soybean Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose intravenous fat emulsion (Experimental): Subjects in this arm will receive approximately 1 g/kg/d IV of intravenous soybean oil (Intralipid).
  Interventions: Drug: Intralipid
- standard dose intravenous fat emulsion (Active Comparator): Subjects in this arm will receive approximately 3 g/kg/d IV of intravenous soybean oil (Intralipid).
  Interventions: Drug: Intralipid

INTERVENTIONS:
Drug: Intralipid — The subject will receive 1 g/kg/d of the standard intravenous fat emulsion while receiving Parenteral Nutrition until discharge from the hospital, death or 100 days of life, whichever comes first.
  Other Names: soybean oil
  Arms: low dose intravenous fat emulsion
Drug: Intralipid — The subject will receive 3 g/kg/d of the standard intravenous fat emulsion while receiving Parenteral Nutrition until discharge from the hospital, death or 100 days of life, whichever comes first.
  Other Names: soybean oil
  Arms: standard dose intravenous fat emulsion

SUMMARY:
Neonates with congenital/acquired gastrointestinal disorders are at high risk for Parenteral Nutrition Associated Cholestasis (PNAC). Besides enteral nutrition, standard therapies to prevent and treat PNAC have been limited and marginal. Recently, the dose and composition of standard intravenous fat emulsions have implicated in the development and progression of PNAC.

In this study, neonates with congenital/acquired gastrointestinal disorders will be randomized, in a unblinded fashion, to receive either the standard dose of an intravenous omega-6 fatty acid emulsion or a low dose of an intravenous omega-6 fatty acid emulsion throughout their course of PN or until hospital discharge, death or 100 days of life, whichever comes first. The primary outcome will be the presence of cholestasis.

DETAILED DESCRIPTION:
Parenteral Nutrition (PN) acts as an intravenous source of both macronutrients and micronutrients when enteral feeds are not possible. Intravenous fat emulsions often supplement PN and provide a dense source of non-protein calories and essential fatty acids. Although PN is life-sustaining, it is associated with a myriad of life-threatening complications including Parenteral Nutrition Associated Cholestasis (PNAC). Children dependent on PN for an extended period of time are high risk for liver failure.

The etiology of PNAC remains poorly understood. Neonates with congenital and acquired gastrointestinal disorders are at high risk for PNAC and its subsequent complications. Examples of these gastrointestinal disorders include gastroschisis, volvulus, atresias, dysmotility and malabsorption disorders, pseudo-obstruction, and Hirschsprung's disease. These disorders often render the gut non-functional for extended periods of time. As a result, these patients become PN-dependent and develop PNAC.

Specific PN components have been implicated in the pathogenesis of PNAC. More recently, standard intravenous fat emulsions have been labeled as one of the main culprits contributing to PNAC. Standard intravenous fat emulsions are dosed as high as 4 g/kg/d and are derived from soybean and/or safflower oil, which are rich in omega-6 fatty acids and phytosterols and contain a paucity of omega-3 fatty acids. It is unclear if the dose or high omega-6 fatty acid:omega-3 fatty acid ratio and phytosterols is responsible for the development of PNAC.

The primary specific aim of this study is to determine if PNAC is related to the amount of standard intravenous fat emulsion administered to neonates with congenital/acquired gastrointestinal disorders. The investigators hypothesize that the PNAC is unrelated to the dose of intravenous fat emulsions. To test this hypothesis, neonates with congenital/acquired gastrointestinal disorders will be randomized to low dose standard soybean based parenteral fat, 1 g/kg/d, or standard dose soybean parenteral fat, 3 g/kg/d. Secondary outcomes include: mortality rate, length of stay, and anthropometric measurements at 28 days of life and at the end of the hospital stay, which is expected to be an average of 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* congenital or acquired gastrointestinal disorder
* age less than 5 days of life

Exclusion Criteria:

* congenital intrauterine infection know to be associated with liver involvement
* known structural liver abnormalities
* known genetic disorders (trisomy 21, 13, and 18)
* inborn errors of metabolism
* infants meeting the criteria for terminal illness (ph:6.8>2 hours)

Ages: 1 Minute to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Calkins, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Saint Louis University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 subjects were enrolled in the study. Only subjects who required > 14 days of parenteral nutrition and who had an abdominal surgery were included in the final analysis.
Period: Overall Study
Arm/Group | Low Dose Intravenous Fat Emulsion | Standard Dose Intravenous Fat Emulsion
Started | 20 | 16
Completed | 20 | 15
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Intravenous Fat Emulsion | Standard Dose Intravenous Fat Emulsion | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Continuous [Mean (Standard Deviation); unit: days] | 1.3 (1.4) | 1.3 (1.1) | 1.3 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 18
  Not Hispanic or Latino | 13 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 17 | 14 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Presence of Cholestasis
Description: Cholestasis will be defined by a direct bilirubin > 2 mg/dL
Time Frame: prior to 100 days of life, hospital discharge, or death whichever comes first
Measure: Number; unit: participants
Arm/Group | Low Dose Intravenous Fat Emulsion | Standard Dose Intravenous Fat Emulsion
Number analyzed (Participants) | 20 | 16
participants
  Presence of Cholestasis-Yes | 6 | 6
  Presence of Cholestasis-No | 14 | 10

2. Secondary Outcome: Mortality Rate
Description: death
Time Frame: at the end of the hospital stay which is expected to be an average of 5 weeks
Measure: Number; unit: participants
Arm/Group | Low Dose Intravenous Fat Emulsion | Standard Dose Intravenous Fat Emulsion
Number analyzed (Participants) | 20 | 16
participants | 0 | 0

3. Secondary Outcome: Anthropometric Measurements
Description: Growth will be assessed by growth velocity at 28 days of age
Time Frame: 28 days of age
Measure: Mean (Standard Deviation); unit: g/d
Arm/Group | Low Dose Intravenous Fat Emulsion | Standard Dose Intravenous Fat Emulsion
Number analyzed (Participants) | 20 | 16
g/d | 18 (8) | 24 (16)

4. Secondary Outcome: Anthropometric Measurements
Description: Growth will be assessed by weight at the time of hospital discharge (approximately 5 weeks)
Time Frame: approximately 5 weeks
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Low Dose Intravenous Fat Emulsion | Standard Dose Intravenous Fat Emulsion
Number analyzed (Participants) | 20 | 16
g | 3.4 (0.9) | 3.5 (0.7)

ADVERSE EVENTS:
Time Frame: Til hospital discharge, which is an average of approximately 5 weeks
Arm/Group | Low Dose Intravenous Fat Emulsion | Standard Dose Intravenous Fat Emulsion
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/16
Other Adverse Events (participants affected / at risk) | 0/20 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Intravenous Fat Emulsion (N=20) | Standard Dose Intravenous Fat Emulsion (N=16)
hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No